CLINICAL TRIAL: NCT05833113
Title: Effects of Transcutaneous Electrical Nerve Stimulation for Postoperative Quality of Recovery After Shoulder Surgery: A Randomized Controlled Trial
Brief Title: Effects of Transcutaneous Electrical Nerve Stimulation for Postoperative Quality of Recovery After Shoulder Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karaman Training and Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 03-2023/15
Record Dates: First submitted 2023-04-17; First posted 2023-04-27 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2023-04

CONDITIONS: Quality of Recovery
Keywords: Interscalene brachial plexus block; Transcutaneous electrical nerve stimulation; Rebound pain
MeSH Terms: interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gruop Control (Placebo Comparator): The patients will be received an ultrasound-guided interscalene brachial plexus block and postoperative Placebo-TENS applied.
  Interventions: Device: Placebo-Transcutaneous Electrical Nerve Stimulation (TENS)
- Group TENS (Active Comparator): The patients will be received an ultrasound-guided interscalene brachial plexus block and postoperative TENS applied.
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation (TENS)

INTERVENTIONS:
Device: Placebo-Transcutaneous Electrical Nerve Stimulation (TENS) — Patients will receive 2 mg midazolam and 50 ug fentanyl for sedation before the block procedure. Each patient will be positioned appropriately, then a high-frequency linear array transducer (13-6 MHz) will be placed in the interscalene region to define the brachial plexus on the short axis. Under sterile conditions, 50 mm block needle will be advanced through the interscalene groove. After localization and negative aspiration, 15 ML of 5% bupivacaine drug will be injected into the interscalene area.
  The control group will also receive the TENS-pants electrodes, connected to TENS treatment. In the placebo-TENS applications on the painful area, 2 channels with 4 electrodes in the acute period will be applied. However, the TENS treatment to the control group will be set so that no electricity will reach the patient.
  A multimodal analgesia regimen will be applied postoperatively
  Arms: Gruop Control
Device: Transcutaneous Electrical Nerve Stimulation (TENS) — Patients will receive 2 mg midazolam and 50 ug fentanyl for sedation before the block procedure. Each patient will be positioned appropriately, then a high-frequency linear array transducer (13-6 MHz) will be placed in the interscalene region to define the brachial plexus on the short axis. Under sterile conditions, 50 mm block needle will be advanced through the interscalene groove. After localization and negative aspiration, 15 ML of 5% bupivacaine drug will be injected into the interscalene area.
  In the TENS applications on the painful area, 2 channels with 4 electrodes in the acute period will be applied. TENS device will be applied 4 times a day with treatment periods of 30 minutes.
  A multimodal analgesia regimen will be applied postoperatively
  Arms: Group TENS

SUMMARY:
Transcutaneous Electrical Nerve Stimulation (TENS) has been reported to reduce postoperative pain scores and opioid consumption after postoperative. This study aims to evaluate the effect of TENS application on recovery quality after interscalene block for shoulder surgery.

DETAILED DESCRIPTION:
Shoulder rotator cuff repair and acromioplasty are associated with severe pain after surgery. Interscalene block (ISB) is the gold standard for shoulder surgery, but the block duration does not exceed 6-8 hours. In addition, after the resolution of ISB, patients experience severe pain and need high doses of opioids. Rebound pain is observed in the postoperative period after the effect of the nerve block abolition. Rebound pain affects the quality of recovery and sleep quality in postoperative.

Transcutaneous Electrical Nerve Stimulation (TENS) is a method of pain relief that uses cutaneously applied electrodes for delivering electrical signals to peripheral nerves through the intact skin. TENS is safe and effective for acute postoperative pain treatment. In addition, TENS has been used in anesthesia to treat postoperative nausea vomiting, and labor analgesia beyond providing analgesia.

We hypothesized that TENS application would reduce the incidence of rebound pain, reduce the need for postoperative opioids, and improve recovery and sleep quality.

This study will be conducted as a single-center, prospective, randomized, double-blinded trial in a university hospital. Patients scheduled for elective shoulder surgery will be screened for enrollment in the study.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing shoulder surgery
* Having signed a written informed consent form,
* ASAI-III

Exclusion Criteria:

* Inadequate indication for interscalene block (Coagulation disorder, local infection of block site, Diaphragmatic paralysis, Allergy to local anesthetics)
* Neuropathic disorder
* Severe cardiopulmonary disease
* Systemic steroid use
* Chronic opioids use
* Ucontrolled Diabetes
* Psychiatric disorders,
* Pregnancy,
* Severe obesity (body mass index > 35 kg/m2)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-04-27 (Actual); Primary Completion 2024-03-10 (Actual); Study Completion 2024-03-24 (Actual)

PRIMARY OUTCOMES:
Quality of Recovery-15 score | Postoperative 24th hour
  Minimum value: 0, Maximum value: 150, higher scores mean better.

SECONDARY OUTCOMES:
Quality of Recovery-15 score | postoperative day 2 and 7
  Minimum value: 0, Maximum value: 150, higher scores mean better.
Numerical Rating Scale | 48 hours
  Range 0-10, 0=no pain, 10=the worse pain ever.
Opioid consumption | 48 hours
  Opioid consumption
The difference of pain score before and after interscalene block resolution | First 24 hours after interscalene block effect disappears
  The difference in the pain score between when the block is working and when it has resolved. Pain scores (0 = no pain; 10 = worst pain imaginable) using a Numerical Rating Scale (NRS) ranging from 0 to 10.
Incidence of rebound pain | 24 hours after surgery
  Rebound pain is described as severe pain (NRS ≥ 7)
Sleep Quality measured with Likert Scale | One week after surgery
  Patients' perceived sleep quality will be assessed with a Likert scale. Likert scale is scored from Likert scale where 1 = very dissatisfied, 2 = dissatisfied, 3 = neutral, 4 = satisfied and 5 = very satisfied.
Number of Participants with Surgical infection | Postoperative 14 days
  Number of Participants diagnosed with surgical infection

CONTACTS AND LOCATIONS:
Locations (1):
- Karaman Training and Research Hospital, Karaman, Turkey (Türkiye)